CLINICAL TRIAL: NCT00941733
Title: Randomized Study of IN.PACT Amphirion™ Drug Eluting Balloon vs. Standard PTA (Percutaneous Transluminal Angioplasty) for the Treatment of Below the Knee Critical Limb Ischemia
Brief Title: Study of IN.PACT Amphirion™ Drug Eluting Balloon vs. Standard PTA for the Treatment of Below the Knee Critical Limb Ischemia
Acronym: INPACT-DEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P998
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Critical Lower Limb Ischemia
Keywords: BTK; CLI; PTA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Eluting Balloon (Experimental): Intervention: IN.PACT Amphirion™
  Interventions: Device: IN.PACT Amphirion
- Standard PTA (Active Comparator): Intervention: Standard PTA
  Interventions: Device: Standard PTA

INTERVENTIONS:
Device: IN.PACT Amphirion — Balloon Angioplasty
  Arms: Drug Eluting Balloon
Device: Standard PTA — Balloon Angioplasty
  Arms: Standard PTA

SUMMARY:
This is a prospective, multi-center, randomized (2:1) trial of symptomatic patients with critical limb ischemia (CLI) secondary to atherosclerotic lesions (stenotic or occluded) of the infrapopliteal vessels. Patients will undergo a percutaneous transluminal endovascular procedure with either the IN.PACT Amphirion™ drug eluting balloon or with a standard (Percutaneous Transluminal Angioplasty) PTA balloon. Patients will be followed with pre-study, post-study, and follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Age ≥18 years and ≤85 years
* Patient or patient's legal representative have been informed of the nature of the study, agrees to participate and has signed an Ethical Committee approved consent form
* Female patients of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation
* Patient has documented chronic Critical Limb Ischemia (CLI) in the target limb prior to the study procedure with Rutherford Category 4, 5 or 6
* Life expectancy >1 year in the Investigator's opinion

General Angiographic Inclusion Criteria

* Reference vessel(s) diameter between 2 and 4 mm
* Single or multiple lesions with ≥70% diameter stenosis (DS) of different lengths in one or more main afferent crural vessels including the tibioperoneal trunk
* At least one non occluded crural vessel with angiographically documented run-off to the foot either direct or through collaterals

Angiographic Inclusion Criteria for Late Lumen Loss (LLL) assessment

* Angio-target lesion (TL) is one identifiable single solitary or series of multiple adjacent lesions with a diameter stenosis (DS) ≥70% and a cumulative length ≤100 mm that can be covered by a single IN.PACT Amphirion™ (10 mm balloon landing zone in both edges is mandatory)
* Angio-target lesion (TL) is the only lesion in that vessel (only one Angio-TL per patient is allowed)

Exclusion Criteria:

General Exclusion Criteria

* Patient unwilling or unlikely to comply with Follow-Up schedule
* Planned major index limb amputation

General Angiographic Exclusion Criteria

* Lesion and / or occlusions located or extending in the popliteal artery or below the ankle joint space
* Inflow lesion or occlusion in the ipsilateral Iliac, Superficial Femoral Artery (SFA), popliteal arteries with length ≥15 cm
* Significant (≥50% DS) inflow lesion or occlusion in the ipsilateral Iliac, Superficial Femoral Artery (SFA) and popliteal arteries left untreated
* Previously implanted stent in the target lesions(s)
* Aneurysm in the target vessel
* Acute thrombus in the target limb

General Procedural Exclusion Criteria

* Failure to obtain a <30% residual stenosis in pre-existing, hemodynamically significant (≥50% diameter stenosis (DS) and <15 cm length) inflow lesions in the ipsilateral iliac, SFA and popliteal artery. No Drug Eluting Stents (DES) and / or Drug Eluting Balloon (DEB) allowed for the treatment of inflow lesions.
* Failure to cross the TL with a 0.014" guide wire
* Use of alternative therapy, e.g. atherectomy, cutting balloon, laser, radiation therapy, DES as part of the index procedure

ANGIOGRAPHIC cohort General Exclusion Criteria:

- Glomerular Filtration Rate (GFR) <30 ml/min except for patients with renal end stage disease on chronic haemodialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Heart Center Leipzig - University Hospital; Thomas Zeller, MD, Principal Investigator — University Heart Center Freiburg - Bad Krozingen; Iris Baumgartner, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (13):
- Medical University Graz, Graz, Austria
- Belgium (4):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - ZOL St. Jan, Genk
  - Ghent University Hospital, Ghent
- Germany (4):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Medical Care Center, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Park-Krankenhaus Leipzig, Leipzig
- Villa Maria Eleonora Hospital, Palermo, Italy
- St. Antonius Hospital, Nieuwegein, Netherlands
- Switzerland (2):
  - University of Bern, Bern
  - Luzerner Kantonsspital, Lucerne

REFERENCES:
- [Derived] Zeller T, Micari A, Scheinert D, Baumgartner I, Bosiers M, Vermassen FEG, Banyai M, Shishehbor MH, Wang H, Brodmann M; IN.PACT DEEP Trial Investigators. The IN.PACT DEEP Clinical Drug-Coated Balloon Trial: 5-Year Outcomes. JACC Cardiovasc Interv. 2020 Feb 24;13(4):431-443. doi: 10.1016/j.jcin.2019.10.059. PMID 32081236
- [Derived] Zeller T, Baumgartner I, Scheinert D, Brodmann M, Bosiers M, Micari A, Peeters P, Vermassen F, Landini M, Snead DB, Kent KC, Rocha-Singh KJ; IN.PACT DEEP Trial Investigators. Drug-eluting balloon versus standard balloon angioplasty for infrapopliteal arterial revascularization in critical limb ischemia: 12-month results from the IN.PACT DEEP randomized trial. J Am Coll Cardiol. 2014 Oct 14;64(15):1568-76. doi: 10.1016/j.jacc.2014.06.1198. PMID 25301459
- [Derived] Zeller T, Baumgartner I, Scheinert D, Brodmann M, Bosiers M, Micari A, Peeters P, Vermassen F, Landini M; IN.PACT DEEP Trial Investigators. IN.PACT Amphirion paclitaxel eluting balloon versus standard percutaneous transluminal angioplasty for infrapopliteal revascularization of critical limb ischemia: rationale and protocol for an ongoing randomized controlled trial. Trials. 2014 Feb 19;15:63. doi: 10.1186/1745-6215-15-63. PMID 24552184
- See also: Zeller et al. Drug-Eluting Balloon Versus Standard Balloon Angioplasty for Infrapoplliteal Arterial Revascularization in CLI - 12-Month Results from the IN.PACT DEEP Randomized trial.Journal of the American College of Cardiology 2014; 64; 15 — http://www.ncbi.nlm.nih.gov/pubmed/24552184

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard PTA: Standard PTA balloon: Balloon Angioplasty
Period: Overall Study
Arm/Group | Drug Eluting Balloon | Standard PTA
Started | 239 | 119
Completed | 165 (1 year follow-up) | 91 (1 year follow-up)
Not Completed | 74 | 28
Not completed — Death | 24 | 10
Not completed — Withdrawal by Subject | 14 | 6
Not completed — Adverse Event | 20 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 15 | 6

BASELINE CHARACTERISTICS:
Population: The total sample size for the study was planned to be 357 subjects, which was intended to fully power the trial for the endpoints of LLL and the composite safety endpoint based on initial estimates of event rates and effect sizes. The endpoint of 12-month TLR was powered to 65% with the indicated sample size.
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Eluting Balloon | Standard PTA | Total
Number analyzed (Participants) | 239 | 119 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (8.2) | 71.7 (9.9) | 72.5 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 35 | 92
  Male | 182 | 84 | 266
Region of Enrollment [Number; unit: participants]
  Germany | 73 | 35 | 108
  Switzerland | 31 | 15 | 46
  Belgium | 60 | 31 | 91
  Austria | 47 | 25 | 72
  Italy | 26 | 13 | 39
  Netherlands | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Late Lumen Loss (LLL) of the Target Lesion by Quantitative Vascular Angiography (QVA)
Description: The difference between minimum lumen diameter (MLD) immediately after Percutaneous Transluminal Angioplasty (PTA) and MLD at 12 months follow-up
Time Frame: 12 months or at Target Lesion Revascularization (TLR) time
Population: ITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 239 | 119
mm | 0.605 (0,775) | 0.616 (0.781)

2. Primary Outcome: Clinically Driven Target Lesion Revascularization (TLR) of the Target Lesion in the Amputation Free Surviving Patients
Description: Percentage of participants in the amputation free survival population with Clinically driven Target Lesion Revascularization (CD-TLR) at 12 months, CD-TLR defined as any TLR of the target lesion associated with Deterioration of Rutherford Class and / or increase in size of pre-existing wounds and / or occurrence of a new wound(s).
Time Frame: 12 months
Population: Amputation free surviving meaning participants without an amputation at 12 months. This analysis population consists of 196 participants in the Drug Eluting Balloon arm and 107 participants in the Standard PTA arm.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 196 | 107
percentage of participants analyzed | 9.2 | 13.1

3. Primary Outcome: Composite of All Cause Death, Major Amputation and Clinically Driven Target Lesion Revascularization (CD-TLR)
Description: Percentage of participants experiencing all cause death, major amputation and clinically driven Target Lesion Revascularization (CD-TLR) at 6 months. CD-TLR defined as any TLR of the target lesion associated with Deterioration of Rutherford Class and / or increase in size of pre-existing wounds and / or occurrence of a new wound(s)
Time Frame: 6 months
Population: Percentage based on number of evaluable subjects for safety events (232 participants in the drug eluting balloon arm and 114 patients in the Standard PTA arm). All randomized subjects experiencing at least one component for the safety endpoint or with follow-up of at least 330 days post-procedure.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 232 | 114
percentage of participants analyzed | 17.67 | 15.79

4. Secondary Outcome: Amputation Free Survival
Description: Percentage of participants with a 1 year amputation free survival.
Time Frame: 12 months
Population: Percentage based on number of evaluable subjects for safety events (227 participants in the drug eluting balloon arm and 111 patients in the Standard PTA arm). All randomized subjects experiencing at least one component for the safety endpoint or with follow-up of at least 330 days post-procedure.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 227 | 111
percentage of participants analyzed | 81.1 | 89.2

5. Secondary Outcome: Rate of Wound Healing
Description: Percentage of participants with completed wound healing, wound healing as defined as core lab adjudication of > 50% area/volume reduction of baseline ulcer(s) in the treated leg at 1 year.
Time Frame: 12 months
Population: Patients with pre-existing wounds and/or occurence of new wounds
Measure: Number; unit: percentage of patients analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 164 | 91
percentage of patients analyzed | 73.8 | 76.9

6. Secondary Outcome: Amputation Free Survival and Wound Healing
Description: Percentage of participants with a 1 year amputation free survival and wound healing. Wound healing is defined as core lab adjudication of > 50% area/volume reduction of baseline ulcer(s) in the treated leg at a specified time point.
Time Frame: 12 months
Population: Percentage based on number of evaluable subjects for safety events (206 participants in the drug eluting balloon arm and 103 patients in the Standard PTA arm). All randomized subjects experiencing at least one component for the safety endpoint or with follow-up of at least 330 days post-procedure.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 206 | 103
percentage of participants analyzed | 58.7 | 68.0

7. Secondary Outcome: Amputation Free Survival and Resolved Critical Limb Ischemia (CLI)
Description: Percentage of participants with an amputation free survival and resolved Critical Limb Ischemia (CLI) at 1 year.
Time Frame: 12 months
Population: Percentage based on number of evaluable subjects for safety events (205 participants in the drug eluting balloon arm and 103 patients in the Standard PTA arm). All randomized subjects experiencing at least one component for the safety endpoint or with follow-up of at least 330 days post-procedure.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 205 | 103
percentage of participants analyzed | 57.1 | 66.0

8. Secondary Outcome: Death, Amputation and Clinically Driven Target Lesion Revascularization (TLR)
Description: Percentage of participants that experienced death, amputation and clinically driven Target Lesion Revascularization (TLR) at 1 year.
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 227 | 111
percentage of participants analyzed | 39.6 | 34.2

9. Secondary Outcome: Primary Sustained Clinical Improvement
Description: Percentage of participants that experienced primary sustained clinical improvement at 1 year, specified as an improvement shift in the Rutherford classification of one class in amputation free, clinically driven target lesion revascularization (TLR) free surviving subjects.
Time Frame: 12 months
Population: Analysis population consists of amputation free, clinically driven (target lesion revascularization)TLR free surviving subjects
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 163 | 91
percentage of participants analyzed | 69.3 | 68.1

10. Secondary Outcome: Secondary Sustained Clinical Improvement
Description: Percentage of participants that experienced a secondary sustained clinical improvement, specified as an improvement shift in the Rutherford classification of one class including the need for clinically driven TLR in amputation free surviving subjects at 1 year.
Time Frame: 12 months
Population: as for outcome 9
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 163 | 91
percentage of participants analyzed | 73.6 | 78.0

11. Secondary Outcome: Quality of Life Assessment by EQ5D
Description: Quality of life assessment by EQ5D at 1 year compared to baseline. EQ-5D is a standardised measure of health status and economic appraisal. The EQ-5D-3L essentially consists of 2 parts:the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: (1) no problems, (2) some problems, (3) extreme problems. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
  EQ-5D health states can be converted into a single summary index where 0.0='worst possible outcome' and 1.0='best possible outcome'.
Time Frame: 12 months
Population: Effectiveness Analysis sets - all randomized subjects with available data for EQ5D at baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 157 | 91
units on a scale | 0.6975 (0.3080) | 0.7445 (0.3035)

12. Secondary Outcome: Walking Capacity Assessment
Description: Walking Impairment assessment by WIQ at 1 year compared to baseline. The Walking Impairment Questionnaire (WIQ) is a questionnaire for evaluating walking impairment in patients with peripheral arterial disease (PAD). This can be used to identify patients with significant impairment and to monitor effectiveness of therapeutic interventions. The questionnaire was self-administered by the patients and contains three domains measuring three important factors of walking impairment in patients with intermittent claudication: (1) difficulty walking a distance during the past month, (2) difficulty walking at a certain speed during the past month, (3) symptoms associated with walking impairment. For each separate domain, a subscore was calculated. The total WIQ score was defined as the mean of the three subscores.
  A WIQ score of 42.5 or less identified low performers; while a score of 75.5 or more identified high performers. The WIQ score range is 0 (minimum) - 100 (maximum).
Time Frame: 12 months
Population: Effectiveness Analysis sets - all randomized subjects with available data for Walking Impairment assessment at baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 76 | 38
units on a scale | 74.6 (35.2) | 75.4 (31.7)

13. Secondary Outcome: MAE (Major Adverse Events)
Description: Percentage of participants with a MAE (Major Adverse Events) at 1 year. Major Adverse Events, defined as Death of any Cause, Major Amputation of target limb, Minor Amputation of target limb
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 227 | 111
percentage of participants analyzed | 35.2 | 25.2

14. Secondary Outcome: Device Success
Description: Percentage of device success defined as exact deployment of the device according to the instructions for use as documented with suitable imaging modalities
Time Frame: Day 1
Population: Number of device deployments
Measure: Number; unit: percentage of device deployments
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 355 | 189
percentage of device deployments | 98.0 | 96.3

15. Secondary Outcome: Technical Success
Description: Percentage of technical success defined as successful vascular access and completion of the endovascular procedure and immediate morphological success with less or equal to 50% residual diameter reduction of the treated lesion on completion angiography
Time Frame: Day 1
Population: Number of device deployments
Measure: Number; unit: percentage of device deployments
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 355 | 189
percentage of device deployments | 93.2 | 88.4

16. Secondary Outcome: Procedural Success
Description: Percentage of patients with a procedural success defined as combination of technical success, device success and absence of procedural complications
Time Frame: Day 1
Population: All randomized subjects with available data
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 238 | 119
percentage of participants analyzed | 98.3 | 100

17. Secondary Outcome: Days of Hospitalization
Description: Days of hospitalization at 1 year
Time Frame: 12 months
Population: All randomized subjects with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 238 | 119
days | 4.5 (8.5) | 4.0 (7.2)

18. Secondary Outcome: Improvement % Diameter Stenosis (%DS) of the Target Leasion (TL) Assessed by Quantitative Vascular Angiography (QVA)
Description: Percentage of participants with an improvement in percent diameter stenosis (%DS) of the target leasion (TL) assessed by Quantitative Vascular Angiography (QVA)
Time Frame: 12 months
Population: Angiographic subgroup only. Angio-target lesion is one identifiable single solitary or series of multiple adjacent lesions with a diameter stenosis higher than 70% and a cumulative length less than 100 mm that can be covered by a single IN.PACT Amphirion™; and Angio-target lesion is the only lesion in that vessel.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Drug Eluting Balloon | Standard PTA
Number analyzed (Participants) | 61 | 31
percentage of participants analyzed | 82.0 | 71.0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Drug Eluting Balloon | Standard PTA
Serious Adverse Events (participants affected / at risk) | 197/239 | 92/119
Other Adverse Events (participants affected / at risk) | 220/239 | 108/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Eluting Balloon (N=239) | Standard PTA (N=119)
Anaemia (Blood and lymphatic system disorders) | 10 (12) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 4 (4)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac failure (Cardiac disorders) | 24 (32) | 10 (11)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (4) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Heart valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 7 (8) | 2 (2)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (2)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 2 (2)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 2 (3)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site rash (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 7 (11) | 2 (2)
Death (General disorders) | 4 (4) | 2 (2)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 3 (4) | 0 (0)
Impaired healing (General disorders) | 28 (36) | 9 (13)
Inflammation (General disorders) | 2 (2) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 2 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 0 (0)
Pain (General disorders) | 2 (3) | 5 (5)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (5) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (2)
Erysipelas (Infections and infestations) | 3 (3) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 13 (15) | 7 (7)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 10 (10) | 4 (4)
Intervertebral discitis (Infections and infestations) | 1 (1) | 3 (3)
Localised infection (Infections and infestations) | 7 (11) | 5 (5)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 7 (8) | 2 (2)
Pneumonia (Infections and infestations) | 7 (8) | 4 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (4) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 12 (12) | 8 (16)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 8 (10) | 2 (3)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriogram coronary abnormal (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Blood glucose fluctuation (Investigations) | 2 (2) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
White blood cell count (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 10 (10) | 2 (3)
Cerebrovascular stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (5) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (6) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 (10) | 2 (3)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 3 (3) | 2 (2)
Angioplasty (Surgical and medical procedures) | 2 (2) | 1 (1)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous shunt operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 2 (2) | 1 (1)
Dialysis device insertion (Surgical and medical procedures) | 0 (0) | 2 (2)
Hospitalisation (Surgical and medical procedures) | 2 (2) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (2) | 0 (0)
Leg amputation (Surgical and medical procedures) | 5 (5) | 0 (0)
Nail operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral revascularisation (Surgical and medical procedures) | 12 (25) | 7 (9)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 7 (7) | 2 (2)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Arterial spasm (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis limb (Vascular disorders) | 21 (25) | 11 (14)
Arterial thrombosis limb (Vascular disorders) | 3 (3) | 2 (5)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 21 (28) | 4 (5)
Femoral arterial stenosis (Vascular disorders) | 19 (28) | 4 (6)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (4) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 6 (6) | 1 (3)
Necrosis ischaemic (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 42 (64) | 22 (59)
Peripheral artery aneurysm (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 2 (2)
Peripheral embolism (Vascular disorders) | 3 (3) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 2 (2)
Reperfusion injury (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Eluting Balloon (N=239) | Standard PTA (N=119)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (6) | 3 (4)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Hyalosis asteroid (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (3) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Device breakage (General disorders) | 1 (1) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 11 (12) | 8 (10)
Inflammation (General disorders) | 2 (2) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 2 (2)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 6 (6) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 6 (6) | 4 (4)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 6 (6) | 5 (5)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 3 (3)
Paronychia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 5 (5) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 6 (7)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Psychosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 13 (17) | 6 (6)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Angiogram (Investigations) | 2 (2) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol abnormal (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 2 (2)
Blood creatine increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Blood glucose fluctuation (Investigations) | 2 (2) | 2 (2)
Blood glucose increased (Investigations) | 2 (2) | 3 (3)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0)
Scan myocardial perfusion (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign spleen tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 5 (5) | 4 (4)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 11 (13) | 4 (4)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 2 (2) | 0 (0)
Bile duct stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral revascularisation (Surgical and medical procedures) | 6 (7) | 5 (6)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Arterial spasm (Vascular disorders) | 18 (22) | 5 (6)
Arterial stenosis limb (Vascular disorders) | 16 (17) | 5 (6)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Artery dissection (Vascular disorders) | 7 (8) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 10 (10) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 7 (8) | 6 (7)
Haematoma (Vascular disorders) | 9 (9) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 7 (8) | 3 (3)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 4 (4) | 3 (3)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 28 (34) | 11 (14)
Peripheral artery dissection (Vascular disorders) | 3 (3) | 1 (1)
Peripheral embolism (Vascular disorders) | 3 (3) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Vascular shunt (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vessel perforation (Vascular disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days